CLINICAL TRIAL: NCT04684225
Title: Telerehabilitation Approach on Individuals With Hand-Affected Scleroderma
Brief Title: Telerehabilitation on Hand-Affected Scleroderma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Tugba Civi Karaaslan, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISTANBULC2
Record Dates: First submitted 2020-12-19; First posted 2020-12-24 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Scleroderma; Scleroderma, Systemic; Scleroderma Associated Digital Ulcer; Hand Rheumatism; Physiotherapy; Rehabilitation
Keywords: Scleroderma; Systemic sclerosis; Telerehabilitation; Hand therapy
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telerehabilitation (Experimental): Stretching and strengthening exercises, functional exercises, massage techniques, sensory training and breathing exercises will be applied to the patients via telerehabilitation for 3 sessions per week.
  Interventions: Other: Hand Therapy via Telerehabilitation
- Home-exercises (Experimental): Stretching and strengthening exercises, functional exercises, massage techniques, sensory training and breathing exercises will be applied by their own at home for 3 sessions per week.
  Interventions: Other: Hand Therapy via home-exercises
- Control (No Intervention): They will have no intervention for 8 weeks. After the period, they will do home exercises.

INTERVENTIONS:
Other: Hand Therapy via Telerehabilitation — Hand Therapy via Telerehabilitation
  Arms: Telerehabilitation
Other: Hand Therapy via home-exercises — Hand Therapy via home-exercises
  Arms: Home-exercises

SUMMARY:
Telerehabilitation Approach on Individuals with Hand-Affected Scleroderma

DETAILED DESCRIPTION:
The effects of exercises performed by telerehabilitation on individuals with hand-affected scleroderma on range of motion, grip strength, function, sensation, daily life activities and general health will be compared with the effects of home-exercises.

Firstly, the evaluation results will be published; and after all data are collected, the results will be published.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with scleroderma
* Stability of medical treatments
* To be able to adapt to the exercises

Exclusion Criteria:

* The patient has a history of neurological disease or trauma that may affect his symptoms
* Systemic involvement that affects the treatment process
* Being in the active phase of the disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Hand Mobility in Scleroderma (HAMIS) | change from baseline at 8 weeks
  Hand Mobility in Scleroderma is a hand function test developed for adults who have systemic sclerosis. HAMIS consists of 9 items designed to measure all movements assessed in an ordinary range of motion-measured hand test. Each item is graded on a 0-3 scale, where 0 corresponds to normal function and 3 denotes that the individual is unable to perform the item. Each hand is assessed separately. The total score of HAMIS for each hand is 370 Sandqvist and Eklund Vol. 13, No. 6, December 2000 27, which represents a high degree of dysfunction.

SECONDARY OUTCOMES:
9-Hole Peg Test | change from baseline at 8 weeks
  It is used to evaluate patients' hand and finger skills. The pegboard is placed in the middle of the body. It is desirable that 9 wooden pins be placed randomly in the 9-hole wooden block as fast as possible, and then the pins are removed from the wooden block and placed in the storage compartment one by one. These times are measured and recorded with a stopwatch. A total of 20 seconds or more is considered a "loss of skill".
Scleroderma Health Assessment Questionnaire (SHAQ) | change from baseline at 8 weeks
  The Scleroderma Health Assessment Questionnaire is a measurement tool for evaluating function in individuals with systemic scleroderma and has been used in a number of countries. SHAQ is made up of 20 items distributed among eight domains and has five additional domains that assess dysfunctions caused by the symptoms of systemic scleroderma. For this, five visual analogue scales (VASs) are used. The scores on these scales are converted to subscores ranging from 0 to 3 points. The overall score of the questionnaire is the sum of each of the five VAS subscores and the scores for the eight domains, divided by 13. Lower score indicates better health status.
Semmes Weinstein Monofilaman Test | change from baseline at 8 weeks
  The severity of pain and paresthesia symptoms of the patients will be assessed using the 10 cm Visual Analogue Scale. Before the assessment, patients instruct that "0" for "no symptoms", "10" represents "the most severe pain that could be felt" and should mark the point that best describes the symptom. The patient's rest, activity and night pain in the last week will be questioned separately. To evaluate the paresthesia, the most severe paresthesia felt by the patient in the last 1 week will be questioned and it will be asked to mark the place that best expresses paresthesia on the scale. Marked points measure by a ruler and record in centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: TUGBA CIVI KARAASLAN, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Tugba Civi Karaaslan, Istanbul, Buyukcekmece, Cerrahpasa Medical Faculty, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No